CLINICAL TRIAL: NCT02758301
Title: Reveal LINQ™ Heart Failure
Acronym: LINQ HF
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: LINQ HF
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Diagnostic: The Reveal LINQ™ Insertable Cardiac Monitor (ICM) device will be inserted in all subjects for continuous monitoring. After the Reveal LINQ™ device is inserted, the LINQ™ HF investigational RAMware will be downloaded to the LINQ™ ICM.
  Interventions: Device: Reveal LINQ™ Insertable Cardiac Monitor (ICM)

INTERVENTIONS:
Device: Reveal LINQ™ Insertable Cardiac Monitor (ICM) — Insertable Cardiac Monitor with LINQ™ HF Investigational RAMware download

SUMMARY:
The purpose of the LINQ™ HF study is to characterize Reveal LINQ™ derived data from patients with heart failure by assessing the relationship between changes in LINQ™ derived data and other physiologic parameters with subsequent acute decompensated heart failure (ADHF) events.

DETAILED DESCRIPTION:
The study is a prospective, non-randomized, multi-center, observational, pre-market clinical study. The study is expected to be conducted at up to 30 centers in the United States. Up to 300 subjects will be enrolled to achieve approximately 40 heart failure events (no more than two per subject will contribute to the cumulative total). Study subjects will be followed for up to 3 years post-insertion or until official study closure defined as when Medtronic and/or regulatory requirements have been satisfied per the Clinical Investigation Plan and/or by a decision by Medtronic or regulatory authority, whichever occurs first. The expected study duration is approximately 4 years representing 1.5 years of enrollments and 2.5 years of follow-up.

The LINQ™ HF study is a Non-Significant Risk Investigational Device Exemption (IDE) study. The study is utilizing the Reveal LINQ™ device with an investigational LINQ™ HF RAMware download.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient (or patient's legally authorized representative) is willing and able to provide written informed consent
* Patient is willing and able to comply with the protocol, including follow-up visits and CareLink transmissions
* Patient is NYHA Class III, per most recent assessment or at any time within 30 days prior to enrollment
* Patient had a HF event (HF event defined as meeting any one of the following three criteria):

  1. Admission with primary diagnosis of HF within the last 6 months, OR
  2. Intravenous HF therapy (e.g. IV diuretics/vasodilators) or ultrafiltration at any one of the following settings within the last 6 months:

     * Admission with secondary/tertiary diagnosis of HF
     * Emergency Department
     * Ambulance
     * Observation Unit
     * Urgent Care
     * HF/Cardiology Clinic
     * Patient's Home, OR
  3. Patient had the following BNP/NTpro-BNP within the last 3 months: If EF ≥ 50%, then BNP> 200 pg/ml or NTpro-BNP > 400 pg/ml OR If EF <50%, then BNP> 400 pg/ml or NTpro-BNP > 800 pg/ml

Exclusion Criteria:

* Patient is pregnant (all females of child-bearing potential must have a negative pregnancy test within 1 week of enrollment)
* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager
* Patient has severe valvular heart disease as defined by hemodynamically significant valve stenosis and/or prosthetic heart valve
* Patient has existing IPG, ICD, CRT-D or CRT-P device
* Patient has severe renal impairment (eGFR <25mL/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject population for the LINQ™ HF study is patients with heart failure with a NYHA Class III who meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Scripps Green Hospital, La Jolla, California
  - Bay Area Cardiology Associates PA, Brandon, Florida
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Louisiana State University, New Orleans, Louisiana
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Mid America Heart Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Carolinas Medical Center, Charlotte, North Carolina
  - The Lindner Research Center, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Austin Heart PA, Austin, Texas
  - University of Virginia, Charlottesville, Virginia
  - Centra Medical Group Stroobants Cardiovascular Center, Lynchburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reveal LINQ Cohort: Subjects inserted with a Reveal LINQ implantable cardiac monitor
- Enrolled But Not Inserted Group: Subjects who were enrolled in the Reveal LINQ HF study, but did not undergo an insertion attempt of a Reveal LINQ device.
Period: Overall Study
Arm/Group | Reveal LINQ Cohort | Enrolled But Not Inserted Group
Started | 104 | 8
Completed | 70 | 0
Not Completed | 34 | 8
Not completed — Death | 12 | 0
Not completed — Physician Decision | 10 | 1
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lost to Follow-up | 7 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled subjects who underwent an insertion of a Reveal LINQ device
Groups:
- Enrolled But Not Inserted Group: Subjects who were enrolled in the Reveal LINQ HF study, but did not undergo an insertion attempt of a Reveal LINQ device, but had a Baseline Form Completed.
- Total: Total of all reporting groups
Arm/Group | Reveal LINQ Cohort | Enrolled But Not Inserted Group | Total
Number analyzed (Participants) | 104 | 7 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (10.9) | 69.4 (14.7) | 66.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 2 | 69
  Male | 37 | 5 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 101 | 7 | 108
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 1 | 18
  White | 86 | 6 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 104 | 7 | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reveal Device Experiencing an Initial Acute Decompensated Heart Failure (ADHF) Event
Description: A heart failure (HF) event is defined as any cardiovascular-related Health Care Utilizations (HCUs) for any one of the following events.
  * Admission with primary diagnosis of HF
  * Intravenous HF therapy (e.g. IV diuretics/vasodilators) or ultrafiltration at any one of the following settings:
    1. Admission with secondary/tertiary diagnosis of HF
    2. Emergency Department
    3. Ambulance
    4. Observation Unit
    5. Urgent Care
    6. HF/Cardiology Clinic
  Up to 2 ADHF events were intended to be allowed per subject:
  1. One had to be at least 30 days post-Reveal LINQ insertion and is summarized in this section, and
  2. A possible second ADHF event must be greater than 90 days after the first ADHF event
  Only subjects with a LINQ device were included in the analysis, as the goal was to acquire LINQ-collected data leading up to the ADHF event.
Time Frame: 30 days post-Reveal LINQ insertion to 3 years post-implant
Population: Subjects inserted with a Reveal LINQ device
Measure: Number; unit: participants
Arm/Group | Reveal LINQ Cohort | Enrolled But Not Inserted Group
Number analyzed (Participants) | 104 | 0
participants | 36 |

2. Primary Outcome: Number of Participants With a LINQ Device Experiencing a Second Acute Decompensated Heart Failure (ADHF) Events
Description: A heart failure (HF) event is defined as any cardiovascular-related Health Care Utilizations (HCUs) for any one of the following events.
  * Admission with primary diagnosis of HF
  * Intravenous HF therapy (e.g. IV diuretics/vasodilators) or ultrafiltration at any one of the following settings:
    1. Admission with secondary/tertiary diagnosis of HF
    2. Emergency Department
    3. Ambulance
    4. Observation Unit
    5. Urgent Care
    6. HF/Cardiology Clinic
  Up to two ADHF events per subject were intended to be evaluated. The first must be at least 30 days post-Reveal LINQ insertion, and the second, summarized in this section, must be greater than 90 days following the first ADHF event.
  Only subjects with a LINQ device were included in the analysis, as the goal was to acquire LINQ-collected data leading up to the ADHF event.
Time Frame: > 90 days following first Acute Decompensated Heart Failure event to 3 years post-implant
Population: Subjects who experienced an ADHF event at least 30 days post-Reveal LINQ insertion
Measure: Number; unit: participants
Arm/Group | Reveal LINQ Cohort | Enrolled But Not Inserted Group
Number analyzed (Participants) | 36 | 0
participants | 12 |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the period of study consent through device (Reveal LINQ) insertion and throughout follow-up. The last scheduled follow-up visit was 12 months post-device insertion, and then subjects were followed until study closure.
Description: Only adverse events that the study investigators determined were related to the Reveal LINQ system or insertion procedure were collected in this study. Adverse events which were not related to either the Reveal LINQ system or Reveal LINQ insertion procedure were not reported.
Arm/Group | Reveal LINQ Cohort | Enrolled But Not Inserted Group
All-Cause Mortality (participants affected / at risk) | 12/104 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/0
Other Adverse Events (participants affected / at risk) | 0/104 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT02758301/Prot_SAP_000.pdf